CLINICAL TRIAL: NCT04558294
Title: Effect of Ketanserin After LSD Administration on the Acute Response to LSD in Healthy Subjects
Brief Title: Effect of Ketanserin After LSD Administration
Acronym: L-Ket
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: BASEC 2020-00614
Record Dates: First submitted 2020-08-25; First posted 2020-09-22 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-10

CONDITIONS: Healthy
MeSH Terms: interventions — Lysergic Acid Diethylamide; Ketanserin

STUDY DESIGN:
Intervention Model Description: Double-blind, placebo-controlled, random-order 2-period cross-over design with 2 treatment conditions:
  1. 100 μg LSD + ketanserin (40 mg)
  2. 100 μg LSD + placebo
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 100 μg LSD + Ketanserin placebo (Experimental)
  Interventions: Drug: Lysergic Acid Diethylamide; Drug: Ketanserin Placebo
- 100 μg LSD + Ketanserin (40mg) (Experimental)
  Interventions: Drug: Lysergic Acid Diethylamide; Drug: Ketanserin

INTERVENTIONS:
Drug: Lysergic Acid Diethylamide — A moderate dose of 100 μg LSD will be administered.
  Other Names: LSD
Drug: Ketanserin Placebo — Mannitol capsules instead of capsules containing Ketanserin.
  Arms: 100 μg LSD + Ketanserin placebo
Drug: Ketanserin — A dose of 40 mg Ketanserin will be administered.
  Arms: 100 μg LSD + Ketanserin (40mg)

SUMMARY:
LSD (lysergic acid diethylamide) is a serotonergic (5-HT) hallucinogen widely used for recreational and/or ethnomedical purposes. LSD is thought to induce its prototypical psychedelic effects primarily via stimulation of the 5-HT2A receptor. This study investigates whether an LSD experience can be attenuated and shortened using 5-HT2A receptor antagonist ketanserin administration after LSD once the psychedelic effects have established.

DETAILED DESCRIPTION:
LSD is a so-called "classic" or serotonergic hallucinogen or psychedelic.The effects of LSD have been frequently investigated in the past in both healthy participants and patients. In these studies, LSD produced acute transient alterations in waking consciousness including visual perceptual alterations, audio-visual synesthesia, derealization and depersonalization. Moreover, several of these studies described robust and sustained effects of LSD in patients suffering from addiction, anxiety and depression.

Its psychedelic effects are mainly attributed to its potent partial 5-HT2A receptor agonism. Consistently, administration the 5-HT2A receptor antagonist ketanserin (40 mg) prior to the administration of LSD (100 μg) almost completely prevented the acute effects of LSD in another study of our research group (NCT03321136). The present study hypothesis is that ketanserin (40 mg) administered 1h after LSD shortens and reduces the acute subjective effects of LSD (100 μg) compared to LSD alone (100 μg) followed by placebo in healthy humans. Such a finding would confirm a primarily competitive antagonism of ketanserin and LSD at the 5-HT2A receptor in vivo and indicate that LSD produces its psychedelic effects only when present at the receptor.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 25 and 65 years old
2. Sufficient understanding of the German language
3. Understanding of procedures and risks associated with the study
4. Willing to adhere to the protocol and signing of the consent form
5. Willing to refrain from the consumption of illicit psychoactive substances during the study
6. Abstaining from xanthine-based liquids and foods from the evenings prior to the study sessions to the end of the study days
7. Willing not to operate heavy machinery within 48 hours after substance administration
8. Willing to use double-barrier birth control throughout study participation
9. Body mass index between 18-29 kg/m2

Exclusion Criteria:

1. Chronic or acute medical condition
2. Current or previous major psychiatric disorder
3. Psychotic disorder or bipolar disorder in first-degree relatives
4. Hypertension (>140/90 mmHg) or hypotension (SBP<85 mmHg)
5. Hallucinogenic substance use (not including cannabis) more than 20 times or any time within the previous two months
6. Pregnancy or current breastfeeding
7. Participation in another clinical trial (currently or within the last 30 days)
8. Use of medication that may interfere with the effects of the study medication
9. Tobacco smoking (>10 cigarettes/day)
10. Consumption of alcoholic beverages (>20 drinks/week)

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-10-16 (Actual); Primary Completion 2021-08-28 (Actual); Study Completion 2021-09-29 (Actual)

PRIMARY OUTCOMES:
Duration of subjective response | 12 months
  Visual Analog Scales (VAS) will be repeatedly used to assess subjective alterations in consciousness over time. VAS will be presented as 100 mm long horizontal lines marked with "not at all" on the left and "extremely" on the right. The following VAS will be used: "any effect", "good effect", "bad effect", "fear", "stimulated", "nausea", "tiredness", "alteration of hearing", "alteration of vision", "synesthesia", "alteration in sense of time", "the boundaries between myself and my surroundings seemed to blur", "talkative", "open", "trust" and "my focus is directed: outward/inward". Subjects will mark the scale with vertical lines.
Extent of subjective response | 12 months
  Visual Analog Scales (VAS) will be repeatedly used to assess subjective alterations in consciousness over time. VAS will be presented as 100 mm long horizontal lines marked with "not at all" on the left and "extremely" on the right. The following VAS will be used: "any effect", "good effect", "bad effect", "fear", "stimulated", "nausea", "tiredness", "alteration of hearing", "alteration of vision", "synesthesia", "alteration in sense of time", "the boundaries between myself and my surroundings seemed to blur", "talkative", "open", "trust" and "my focus is directed: outward/inward". Subjects will mark the scale with vertical lines.
Plasma concentrations of LSD | 12 months
  LSD plasma concentrations will be measured repeatedly over time using LC-MS/MS techniques (nanogram per milliliter scale).
Plasma concentrations of Ketanserin | 12 months
  LSD plasma concentrations will be measured repeatedly over time using Liquid chromatography-mass spectrometry (LC-MS)/MS techniques (nanogram per milliliter scale).

SECONDARY OUTCOMES:
5 dimensions of altered state of consciousness (5D-ASC) profile total score | 12 months
  Visual analog scale consisting of 94 items. Constructed of five scales and allows assessing mood, anxiety, derealization, depersonalization, changes in perception, auditory alterations, and reduced vigilance. Scales will be presented as 100 mm long horizontal lines marked with vertical lines by the participant.
Adjective mood rating scale (AMRS) | 12 months
  The adjective mood rating scale (AMRS or EWL60S) is a 60-item 4-point Likert scale ("not at all", "somewhat", "rather", "strongly") that allows repeated assessment of mood in 6 dimensions: activation, inactivation, well-being, anxiety/depressed mood, extroversion and introversion, and emotional excitability.The AMRS consists of subscales measuring "activation", "positive mood", "extroversion", "introversion", "inactivation", and "emotional excitability".
States of consciousness questionnaire (SCQ) | 12 months
  This 100-item questionnaire is rated on a 6-point scale (0=none, not at all; 1=so slight cannot decide; 2=slight; 3=moderate; 4=strong (equivalent in degree to any previous strong experience or expectation of this description); 5=extreme (more than ever before in my life and stronger than 4)). Forty-three items embedded into this questionnaire comprise the Mystical Experience Questionnaire (MEQ). The 43 items provide scale scores for each of seven domains of mystical experiences: internal unity (pure awareness, a merging with ultimate reality), external unity (unity of all things, all things are alive, all is one), sense of sacredness (reverence, sacred), noetic quality (encounter with ultimate reality, more real than everyday reality), transcendence of time and space, deeply felt positive mood (joy, peace, love), paradoxicality/ineffability (claim of difficulty in describing the experience in words).
Blood pressure | 12 months
  Repeatedly measured using blood pressure / pulse apparatus (mmHg scale).
Heart rate | 12 months
  Repeatedly measured using blood pressure / pulse apparatus (beats per minute scale).
Body temperature | 12 months
  Repeatedly measured using ear thermometer (degree Celsius scale).
Pupil diameter | 12 months
  Repeatedly measured using pupil distance meter (millimeter scale).
Elliot Humility Scale (EHS) | 12 months
  Assesses the personality trait humility through 13 items on a 5-point Likert scale ranging from "strongly disagree" to "strongly agree".
Jankowski Humility Scale (JHS) | 12 months
  Assesses the personality trait humility through 18 items on a 5-point Likert scale ranging from "not at all" to "strongly".
Arnett Inventory of Sensation Seeking (AISS-d) | 12 months
  Assesses the personality trait of sensation seeking, which is is defined as a need for novel and intense stimulation. It uses 20 items using 4-point scales (1 = "describes me very well" to 4 = "does not describe me at all").
Freiburger Persönlichkeitsinventar (FPI) | 12 months
  The FPI-R version comprises 138 items and covers 12 dimensions of personality: life satisfaction, social orientation, performance orientation, inhibition, excitability, aggressiveness, stress, physical complaints, health concerns, openness, as well as the secondary factors according to Eysenck's Extraversion and Emotionality (Neuroticism). It uses a 2-point scale ("true" and "not true").
Saarbrücker Persönlichkeitsfragebogen (SPF) | 12 months
  The SPF defines empathy as the "reactions of one individual to the observed experiences of another." It assesses 28-items on a 5-point Likert scale ranging from "Does not describe me well" to "Describes me very well". The measure has 4 subscales (Perspective Taking, Fantasy, Empathic Concern, Personal Distress) each made up of 7 different items.
Defense Style Questionnaire (DSQ-40) | 12 months
  The DSQ-40 can provide scores for 20 individual defenses, and scores for the three factors "mature", "neurotic", and "immature". Each item is evaluated on a scale from 1 to 9, where "1" indicates "completely disagree" and "9" indicates "fully agree".

CONTACTS AND LOCATIONS:
Overall Officials: Matthias E Liechti, Dr., MD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- Clinical Pharmacology & Toxicology, University Hospital Basel, Basel, Switzerland

REFERENCES:
- [Derived] Becker AM, Klaiber A, Holze F, Istampoulouoglou I, Duthaler U, Varghese N, Eckert A, Liechti ME. Ketanserin Reverses the Acute Response to LSD in a Randomized, Double-Blind, Placebo-Controlled, Crossover Study in Healthy Participants. Int J Neuropsychopharmacol. 2023 Feb 14;26(2):97-106. doi: 10.1093/ijnp/pyac075. PMID 36342343